CLINICAL TRIAL: NCT07341035
Title: The Effect of Video-Assisted Genital Hygiene Education on Women's Self-Care Agency and Genital Hygiene Behaviors
Brief Title: Genital Hygiene Education on Women's Self-Care Agency and Genital Hygiene Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Banu CİHAN ERDOĞAN, Assistant Professor, Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 06-07-2023/8
Record Dates: First submitted 2025-12-21; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Patient Education; Hygiene; Genital Hygiene
Keywords: women; hygiene; self-care; patient education
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Groups (Experimental): Experimental Group; the women in the experimental group were provided with the relevant forms and asked to complete the Data Collection Form for Women, Self-Care Agency Scale, and Genital Hygiene Behaviors Scale for the pretest. Afterward, they received information about the importance of genital hygiene, key points to consider during genital hygiene, and watched a training video developed by the researchers. This video demonstrated genital hygiene practices on a human model, with the researcher explaining and demonstrating the steps in a practical manner.
  Following the video training, participants completed the same forms again (Data Collection Form for Women, Self-Care Agency Scale, and Genital Hygiene Behaviors Scale) for the midterm test. To assess the long-term effects of the training, the participants were asked to complete the same forms 8 weeks after the training.
  Interventions: Other: Video
- Control Groups (No Intervention): Control Group; the women in the control group were informed about the forms and asked to complete the Data Collection Form for Women, Self-Care Agency Scale, and Genital Hygiene Behaviors Scale for the pretest. They were also informed about the importance of genital hygiene and key points to consider, but no video-assisted training was provided. The control group filled out the same forms for the midterm and posttest assessments, at the same times as the experimental group.

INTERVENTIONS:
Other: Video — The women in the experimental group were provided with the relevant forms and asked to complete the Data Collection Form for Women, Self-Care Agency Scale, and Genital Hygiene Behaviors Scale for the pretest. Afterward, they received information about the importance of genital hygiene, key points to consider during genital hygiene, and watched a training video developed by the researchers. This video demonstrated genital hygiene practices on a human model, with the researcher explaining and demonstrating the steps in a practical manner.
  Following the video training, participants completed the same forms again (Data Collection Form for Women, Self-Care Agency Scale, and Genital Hygiene Behaviors Scale) for the midterm test. To assess the long-term effects of the training, the participants were asked to complete the same forms 8 weeks after the training.
  Arms: Experimental Groups

SUMMARY:
This study aims to examine the effect of video-assisted genital hygiene education on women's self-care agency and genital hygiene behaviors. It is designed as a single-blind, randomized controlled experimental study.

DETAILED DESCRIPTION:
This single-blind, randomized controlled experimental study is designed to assess the impact of video-assisted genital hygiene education on women's self-care agency and genital hygiene behaviors. Participants will be randomly assigned to an intervention group or a control group. Data will be collected using validated self-report instruments at baseline, immediately after the intervention, and during follow-up.

ELIGIBILITY:
* Inclusion Criteria: Patients who were diagnosed with urinary tract infection by a physician, who had no hearing difficulties and visual loss, and who could communicate were included in the study.
* Exclusion Criteria: Patients who were not diagnosed with urinary tract infection, who were hard of hearing, visually impaired, unable to communicate, unable to maintain genital hygiene and who refused to participate in the study were excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 66 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-12-09 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Self-Care Agency Level | Baseline (Pretest, Week 1), immediately after the intervention (Posttest, Week 2), and 3-month follow-up
  Self-care agency will be assessed using the Self-Care Agency Scale, developed by Kearney and Fleischer (1979) and validated in Turkish by Nahcivan (2004).
  The scale consists of 35 items rated on a 5-point Likert scale (0-4), with a total score range of 0 to 140. Higher scores indicate higher levels of self-care agency.
Genital Hygiene Behaviors | Baseline (Pretest, Week 1), immediately after the intervention (Posttest, Week 2), and 3-month follow-up
  Genital hygiene behaviors will be measured using the Genital Hygiene Behaviors Scale, validated by Karahan (2017).
  The scale includes 23 items rated on a 5-point Likert scale (1-5), with total scores ranging from 23 to 115.
  Higher scores indicate more positive genital hygiene behaviors.

CONTACTS AND LOCATIONS:
Locations (1):
- Çankırı Karatekin University, Çankırı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available.

REFERENCES:
- [Background] Dahodwala M, Geransar R, Babion J, de Grood J, Sargious P. The impact of the use of video-based educational interventions on patient outcomes in hospital settings: A scoping review. Patient Educ Couns. 2018 Dec;101(12):2116-2124. doi: 10.1016/j.pec.2018.06.018. Epub 2018 Jun 30. PMID 30087021
- [Background] Massimi A, De Vito C, Brufola I, Corsaro A, Marzuillo C, Migliara G, Rega ML, Ricciardi W, Villari P, Damiani G. Are community-based nurse-led self-management support interventions effective in chronic patients? Results of a systematic review and meta-analysis. PLoS One. 2017 Mar 10;12(3):e0173617. doi: 10.1371/journal.pone.0173617. eCollection 2017. PMID 28282465
- [Background] Mancuso G, Midiri A, Gerace E, Marra M, Zummo S, Biondo C. Urinary Tract Infections: The Current Scenario and Future Prospects. Pathogens. 2023 Apr 20;12(4):623. doi: 10.3390/pathogens12040623. PMID 37111509
- [Background] Cox S, Vleeming M, Giorgi W, Dinant GJ, Cals J, de Bont E. Patients' Experiences, Expectations, Motivations, and Perspectives around Urinary Tract Infection Care in General Practice: A Qualitative Interview Study. Antibiotics (Basel). 2023 Jan 24;12(2):241. doi: 10.3390/antibiotics12020241. PMID 36830152